CLINICAL TRIAL: NCT00538694
Title: A Randomized, Double-Blind, Phase III, Comparative Study of Cidecin™ (Daptomycin) to Rocephin® (Ceftriaxone) in the Treatment of Moderate to Severe Community-Acquired Acute Bacterial Pneumonia Due to S. Pneumoniae
Brief Title: Comparative Study of Cidecin™ (Daptomycin) to Rocephin® (Ceftriaxone) in the Treatment of Moderate to Severe Community-Acquired Acute Bacterial Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: DAP-00-05
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Pneumonia, Bacterial
Keywords: Moderate to severe community-acquired acute bacterial pneumonia due to S. Pneumoniae
MeSH Terms: conditions — Pneumonia, Bacterial | interventions — Daptomycin

INTERVENTIONS:
Drug: daptomycin

SUMMARY:
To evaluate the safety and efficacy of daptomycin in adults who have pneumonia due to Streptococcus pneumoniae.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent.
2. Adults, 18 years of age or older of either gender and of any race. Female patients of childbearing potential MUST be nonpregnant (confirmed by negative serum pregnancy test), nonlactating, and must be willing to practice reliable birth control measures during and for at least 28 days after treatment with study drug(s).
3. Must exhibit clinical signs/symptoms and radiographic appearance of pneumonia: presence of new pulmonary infiltrate on chest radiograph; fever (oral >38.0 degree C/100.4 degree F); and at least one of the following signs and symptoms consistent with the diagnosis of acute bacterial pneumonia: acute onset, chills, chest pain/dyspnea, cough, or sputum production.
4. Pneumonia which: requires hospitalization; requires IV antibiotic therapy; anticipated >=5 days IV therapy; and (for Grade II) O2 saturation <90% and PaO2 <60 mmHg on room air.
5. Provide a suitable sputum specimen for Gram's-stain and culture. If expectorated sputum or transtracheal aspirate: >10 lancet-shaped Gram-positive diplococci/oil-immersion field (1000x); <10 squamous epithelial cells/low-power field (100x); >25 leukocytes/low-power field (100x).
6. An elevated total peripheral white blood cell count (WBC >10,000/mm3); or >15% immature neutrophils (bands), regardless of total peripheral white count; or leukopenia with total WBC <4500/mm3.
7. Willingness to participate in this study and to complete all follow-up assessments.

Exclusion Criteria:

1. Grade I pneumonia risk classification, or Grade II with O2 saturation >90% on room air and/or PaO2 >60 mmHg on room air (based on Fine Score; Attachment 8).
2. Patients with Grade V pneumonia (based on Fine Score; Attachment 8).
3. Respiratory failure without mechanical ventilatory support (i.e., PaO2 / FiO2 <200), or underlying lung disease precluding interpretation of study results (e.g., cystic fibrosis, lung cancer).
4. Loculated empyema.
5. Severe shock (systolic blood pressure <90 mm Hg for >30 minutes not corrected by fluid bolus).
6. Clinical evidence of bacterial meningitis (based on lumbar puncture results).
7. Renal impairment (calculated creatinine clearance <30 mL/min); hepatic dysfunction (ALT/AST more than 3 times the upper limit of normal or bilirubin >=2.0 mg/dL); or clinical or histologic diagnosis of cirrhosis or another form of chronic liver disease, such as chronic active hepatitis.
8. Moribund clinical condition: high likelihood of death during the first 48 hours.
9. Patients who are severely immunocompromised due to underlying disease or exogenous therapies, CD4 counts <100/mm3.
10. Inability to tolerate ceftriaxone or history of allergy to beta-lactam antibiotics (history of rash alone will not exclude a patient).
11. Any individual previously treated with a potentially effective anti-infective agent for >=24 hours immediately prior to enrollment, or prior treatment with any investigational drug (including experimental biologic agents) in previous 30 days or prior therapy with daptomycin.
12. Patients who must continue HMG-CoA reductase inhibitor therapy (e.g., simvastatin, lovastatin, etc) during the study treatment period.
13. Use of >0.5 mg/kg/day prednisone or equivalent for >1 week preceding enrollment.
14. Anticipation that a second systemic antibiotic will be required.
15. Induction chemotherapy within 2 weeks prior to enrollment (or exogenous therapies which are anticipated to result in PMN counts of <200 mm3 during Treatment Phase), or patients with severe neutropenia (<200 PMN cells/mm3).
16. Patients considered unreliable to return for visits or to comply with study procedures.
17. Functionally or surgically asplenic (e.g., sickle cell disease, multiple myeloma).
18. Neoplastic disease, except basal cell or squamous cell cancer of the skin that was active at the time of enrollment or within 1 year prior to enrollment.
19. Women who are pregnant or nursing/lactating.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2000-10-31 (Actual); Primary Completion 2001-09-30 (Actual); Study Completion 2001-09-30 (Actual)

REFERENCES:
- [Result] Pertel PE, Bernardo P, Fogarty C, Matthews P, Northland R, Benvenuto M, Thorne GM, Luperchio SA, Arbeit RD, Alder J. Effects of prior effective therapy on the efficacy of daptomycin and ceftriaxone for the treatment of community-acquired pneumonia. Clin Infect Dis. 2008 Apr 15;46(8):1142-51. doi: 10.1086/533441. PMID 18444848